CLINICAL TRIAL: NCT06928064
Title: Prediction of Postoperative Pain Severity Using Pain Sensitivity Questionnaire Applied in Preoperative Period in Patients Undergoing Breast-Conserving Surgery (Lumpectomy)
Brief Title: Pain Sensitivity Questionnaire Applied in Preoperative Period in Lumpectomy
Acronym: Lumpectomy
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, SEVDE RUMEYSA YILMAZ, medical doctor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: SRYILMAZ; 010.99/16 (Other: Dr Lutfi Kirdar City Hospital)
Record Dates: First submitted 2025-03-20; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Pain Score; Pain Postoperative
Keywords: breast surgery; pain sensivity
MeSH Terms: conditions — Pain, Postoperative | interventions — Preoperative Period; Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Having planned BCS with general anesthesia • Being a female patient between the ages of 18-70: Having planned BCS with general anesthesia Being a female patient between the ages of 18-70 Being evaluated as American Society of Anesthesiologists (ASA) I, II, III Having given written consent to participate in the study
  Interventions: Procedure: Prediction of Postoperative Pain Severity Using Pain Sensitivity Questionnaire Applied in Preoperative Period in Patients Undergoing Breast-Conserving Surgery (Lumpectomy).

INTERVENTIONS:
Procedure: Prediction of Postoperative Pain Severity Using Pain Sensitivity Questionnaire Applied in Preoperative Period in Patients Undergoing Breast-Conserving Surgery (Lumpectomy). — : This study included 74 patients over the age of 18 with American Society of Anesthesiologists (ASA) scores of I, II, or III, who were scheduled to undergo breast-conserving surgery. Ethical approval from the local ethics committee and written informed consent from each patient were obtained. Patient data, including age, ASA score, and comorbidities, were collected, and contact details were recorded for postoperative follow-up.
  The PSQ was administered to all patients during the preoperative period to assess their pain sensitivity. Anesthesia induction and maintenance followed a standardized protocol on the day of surgery. The intraoperative analgesic consumption and the duration of the surgery were documented. Postoperative assessments were conducted 24 hours after the surgery in the general surgery ward, where analgesic use and short pain inventory scores were recorded. Patients were followed up one month postoperatively, and their pain levels were assessed using the Numeric Rating

SUMMARY:
Objective: The Pain Sensitivity Questionnaire (PSQ) is a clinically valuable tool that has been shown to correlate with various experimental pain sensitivity assessments in healthy individuals and patients with chronic pain. In this study, we aimed to investigate the effectiveness of the PSQ in predicting postoperative pain in patients undergoing breast-conserving surgery.

DETAILED DESCRIPTION:
Objective: The Pain Sensitivity Questionnaire (PSQ) is a clinically valuable tool that has been shown to correlate with various experimental pain sensitivity assessments in healthy individuals and patients with chronic pain. In this study, we aimed to investigate the effectiveness of the PSQ in predicting postoperative pain in patients undergoing breast-conserving surgery.

Materials and Methods: This study included 74 patients over the age of 18 with American Society of Anesthesiologists (ASA) scores of I, II, or III, who were scheduled to undergo breast-conserving surgery. Ethical approval from the local ethics committee and written informed consent from each patient were obtained. Patient data, including age, ASA score, and comorbidities, were collected, and contact details were recorded for postoperative follow-up.

The PSQ was administered to all patients during the preoperative period to assess their pain sensitivity. Anesthesia induction and maintenance followed a standardized protocol on the day of surgery. The intraoperative analgesic consumption and the duration of the surgery were documented. Postoperative assessments were conducted 24 hours after the surgery in the general surgery ward, where analgesic use and short pain inventory scores were recorded. Patients were followed up one month postoperatively, and their pain levels were assessed using the Numeric Rating Scale (NRS).

ELIGIBILITY:
Inclusion Criteria:

Having planned BCS with general anesthesia

* Being a female patient between the ages of 18-70
* Being evaluated as American Society of Anesthesiologists (ASA) I, II, III
* Having given written consent to participate in the study

Exclusion Criteria:

Pregnancy

* Being assessed as ASA IV
* Having advanced cardiac, pulmonary and cerebrovascular disease, advanced renal failure, liver failure, history of fentanyl/remifentanyl hypersensitivity, Alzheimer's disease, mental retardation
* Being at a mental level that cannot comply with the evaluations within the scope of the study
* Not having given written consent for any reason

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients between the ages of 18-70 who are scheduled for breast-conserving surgery
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Prediction of Postoperative Pain Severity Using Pain Sensitivity Questionnaire Applied in Preoperative Period in Patients Undergoing Lumpectomy | From March 2024 to August 2024
  This study included 74 patients over the age of 18 with American Society of Anesthesiologists (ASA) scores of I, II, or III, who were scheduled to undergo breast-conserving surgery. Ethical approval from the local ethics committee and written informed consent from each patient were obtained. Patient data, including age, ASA score, and comorbidities, were collected, and contact details were recorded for postoperative follow-up.The aim was to examine the relationship between the PSQ score measured in the preoperative period and the degree of pain in the postoperative period. BPI score and NRS score were used in the evaluation of postoperative pain.

CONTACTS AND LOCATIONS:
Overall Officials: BANU CEVIK, PROFFESSOR, Study Chair — DR LUTFI KIRDAR CITY HOSPİTAL
Locations (1):
- Dr Lutfi Kirdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided